CLINICAL TRIAL: NCT04914572
Title: Using Therapeutic Rainforest Mindful Walking in Generating Positive Mental Well-being Among Undergraduate Students
Brief Title: Therapeutic Rainforest Study in Generating Positive Energy Among Undergraduate Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Goh Yong-Shian, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MindtheGap200
Record Dates: First submitted 2021-06-01; First posted 2021-06-04 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Stress; Anxiety
Keywords: Mental health; well-being; stress;
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: * The first arm of the study includes the use of mindful walking through the therapeutic rainforest trail from Kent Ridge Park to Hort Park and Hort Park back to Kent Ridge Park.
  * The second arm of the study includes a walk through the therapeutic rainforest trail from Kent Ridge Park to Hort Park and Hort Park back to Kent Ridge Park.
  * The third arm of the study includes a walk through the Kent Ridge Road Trail curated by the Office of Facility Management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapeutic rainforest & MIndful walking (Experimental): The first arm uses mindful walking through a 2km forest trail in Singapore. All Interventional and Control arms will conduct their walk between 8 am to 11 am for five occasions weekly. At the T1, participants will attend a Zoom orientation session to familiarize themselves with the route. During this session, participants will need to answer the self-report questionnaire and provide the first saliva sample for the baseline measurement. In T2, a pre-intervention and post-intervention saliva sample will be taken before the walk. This will follow by T3 the following week. At T4, participants will attend a 60 mins reflection session and answer the self-report questionnaire. On T5 and T6, the participants will continue with the therapeutic rainforest mindfulness walk. On T7, a pre-intervention and post-intervention saliva sample will be taken. On T8, participants will attend a 60 mins reflection session and answer the self-report questionnaire.
  Interventions: Other: Therapeutic rainforest mindful walking
- Therapeutic rainforest walk (Experimental): The second arm of the intervention includes walking through a guided forest trail suggested by NParks Board. The collection of samples and answering of the self-report questionnaire will follow the same sequence as the 1st arm of the 3-arm RCT.
  Interventions: Other: Therapeutic rainforest walk
- Campus green walk (Active Comparator): The control for this study includes guided casual walking around the campus green trial conducted at the same intervals as per the interventions. The collection of samples and answering of the self-report questionnaire will also follow the same sequence as the 1 arm of the 3-arm RCT.
  Interventions: Other: Campus Green walk

INTERVENTIONS:
Other: Therapeutic rainforest mindful walking — A two-kilometer trail curated by the National Parks Board, Singapore. The walk will be led by Mindfulness Practitioner who volunteered to be guides for this study.
  Arms: Therapeutic rainforest & MIndful walking
Other: Therapeutic rainforest walk — A two-kilometer trail curated by the National Parks Board, Singapore. The walk will be led by volunteer guides recruited by the research team.
  Arms: Therapeutic rainforest walk
Other: Campus Green walk — A two-kilometer trail curated by the Office of Facility Management, NUS. The walk will be led by volunteer guides recruited by the research team.
  Arms: Campus green walk

SUMMARY:
This study looked into how therapeutic forest walking will impact the well-being of undergraduate students at the National University of Singapore. A three-arm randomized control trial on 108 participants is being planned for this study. The primary aim of this study is to assess the feasibility and primary effect of the Therapeutic Rainforest Walking in generating positive energy among undergraduate students project in enhancing the quality of life, physical, mental, and psycho-social well-being among University students.

ELIGIBILITY:
Inclusion Criteria:

* Current NUS undergraduate students
* No self-reported physical mobility issue
* No self-reported existing mental health conditions
* Enjoys nature

Exclusion Criteria:

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale 4 (PSS-4) | 8 weeks
  4 items, Likert scale (0-lowest, 4-highest) Scoring higher in the scale would translate to higher perceived stress.
Generalised Anxiety Disorder Scale (GAD-7) | 8 weeks
  7 items, Likert scale (0-lowest, 3-highest) Scoring higher in the scale would translate to higher anxiety level.
English Brief Resilience Scale (BRS) | 8 weeks
  6 items, Likert scale (1-lowest, 5-highest) Scoring higher in the scale would translate to higher resilience.
Saliva Cortisol | 8 weeks
  Measured using Passive drool method

CONTACTS AND LOCATIONS:
Overall Officials: Yong Shian Goh, PhD, Principal Investigator — National University of Singapore
Locations (1):
- Alice Lee Centre for Nursing Studies, Singapore, Singapore